CLINICAL TRIAL: NCT02557152
Title: The GentleWave Post-Market Registry
Brief Title: The GentleWave Registry
Status: Completed | Type: Observational
Sponsor: Sonendo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-10
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Root Canal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients that were treated with the GentleWave System
  Interventions: Device: GentleWave System Treatment

INTERVENTIONS:
Device: GentleWave System Treatment

SUMMARY:
The purpose of this registry is to gain a real world perspective for the use and outcomes associated with the Sonendo® GentleWave System usage. The registry population includes up to 500 subjects that have been treated with the Sonendo GentleWave System at up to 25 clinical sites in the United States.

DETAILED DESCRIPTION:
The purpose of this registry is to gain a real world perspective for the use and outcomes associated with the Sonendo® GentleWave System usage.

Up to 25 clinical sites in the United States. Up to 500 subjects that have been treated with the Sonendo GentleWave System. To assess outcomes for teeth treated with the GentleWave System in a commercial setting.

ELIGIBILITY:
Inclusion Criteria:

* One or more teeth treated with the Sonendo GentleWave System

Exclusion Criteria:

* Institutionalized patients or prisoners

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 500 subjects that have been treated with the Sonendo GentleWave System.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Healing | 24 months
  Radiographic analysis and clinical signs and symptoms at 24 months

SECONDARY OUTCOMES:
Retreatment Rates | 24 months
  Rate of retreatment at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim Bradbury, Study Director — Sonendo, Inc.
Locations (3):
- United States (3):
  - Randy Garland, DDS, Encinitas, California
  - SC Endododontics, Santa Ana, California
  - Stacey Woo, DDS, Whittier, California